CLINICAL TRIAL: NCT04510454
Title: Evaluation of a ddPCR Technology for the SARS-CoV-2 Detection in Symptomatic Patients With Suspicion of COVID-19
Acronym: ONCOVID-21
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ONCOVID-21 - ET20-118
Record Dates: First submitted 2020-08-11; First posted 2020-08-12 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Cancer; COVID
Keywords: COVID-19, SARS-CoV-2, ddPCR, cancer, serology
MeSH Terms: conditions — Neoplasms; COVID-19

STUDY DESIGN:
Intervention Model Description: Nasopharyngeal and oropharyngeal samples will be analyzed by the standard RT-qPCR test and the ddPCR assay.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RT-PCR and ddPCR sampling analyses (Experimental): Nasopharyngeal and throat/oropharyngeal swabs analyzed by both RT-PCR and ddPCR
  Interventions: Diagnostic Test: Nasopharyngeal and throat/oropharyngeal swabs analyses by RT-PCR and ddPCR

INTERVENTIONS:
Diagnostic Test: Nasopharyngeal and throat/oropharyngeal swabs analyses by RT-PCR and ddPCR — Nasopharyngeal and throat/oropharyngeal swabs analyzed by both RT-PCR and ddPCR

SUMMARY:
Evaluation of the ddPCR ability to detect the SARS-CoV-2 in nasopharyngeal samples of symptomatic patients with suspected COVID-19 infection using an IgG serological assay (EUROIMMUN Anti-SARS-Cov2 ELISA Ig) as gold/reference standard (FDA validated commercial serologic test).

DETAILED DESCRIPTION:
The Bio-Rad SARS-CoV-2 ddPCR Test is a reverse transcription (RT) droplet digital polymerase chain reaction (ddPCR) test designed to detect RNA from SARS-CoV-2 in specimens (mainly nasopharyngeal, anterior nasal, oropharyngeal and mid-turbinate swab but also nasopharyngeal wash/aspirate and nasal aspirate specimens) collected from individuals who are suspected of COVID-19 infection.

This single assay multiplex test enables a one-well reaction with three sets of the oligonucleotide primers and probes which were reported by CDC. Two were selected from regions of the virus nucleocapsid (N) gene. An additional primer/probe included in the panel is set to detect the human RNase P gene (RP) in control samples and clinical specimens.

RNA isolated and purified from swab specimens is added to the mastermix comprised of reverse transcriptase whereby RNA is converted into cDNA and then amplified, using the Bio-Rad One-Step RT-ddPCR Advanced Kit for Probes.

Briefly, the sample and mastermix RT-ddPCR mixtures are fractionated into up to 20,000 nanoliter-sized droplets in the form of a water-in-oil emulsion. The 96-well RT-ddPCR ready plate containing droplets is sealed with foil using a plate sealer. The emulsions are then thermocycled to achieve reverse transcription to generate cDNA followed by target amplification plus probe hydrolysis in each droplet. After thermocycling is complete, the 96-well RT-ddPCR ready plate is loaded into the Droplet Reader. The Droplet Reader singulates the droplets and flows them past a two-color fluorescence detector (FAM and HEX) in order to determine which contain target (positive) and which do not (negative) for each of the targets identified with the SARS-CoV-2 ddPCR Test: N1, N2 and RP. The ddPCR system uses the QuantaSoft 1.7 and QuantaSoft Analysis Pro 1.0 for analysis software.

ELIGIBILITY:
1. Age ≥ 18 years on the day of signing informed consent.
2. Confirmed diagnosis of any type of solid or hematologic tumor.
3. Ongoing anticancer treatment at the time of inclusion or within the last 3 months prior to inclusion (last treatment administration or last loco regional procedure).
4. Suspicion of COVID-19 infection. Patients must not have underwent diagnostic test and/or chest imaging before inclusion.
5. Covered by a medical/health insurance.
6. Signed and dated IRB/ICE approved informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2021-06-24 (Actual); Study Completion 2021-10-12 (Actual)

PRIMARY OUTCOMES:
To determine the ddPCR ability to detect the SARS-CoV-2 in nasopharyngeal samples of symptomatic patients with suspected COVID-19 infection | At inclusion
  Using IgG serological assay (EUROIMMUN Anti-SARS-Cov2 ELISA Ig) as gold/reference standard (FDA validated commercial serologic test)

SECONDARY OUTCOMES:
To determine the RT-qPCR ability to detect the SARS-CoV-2 in nasopharyngeal samples of symptomatic patients with suspected COVID-19 infection | Third week after inclusion
  Using IgG serological assay (EUROIMMUN Anti-SARS-Cov2 ELISA Ig) as gold/reference standard
To determine the ddPCR and RT-qPCR abilities to detect the SARS-CoV-2 in oropharyngeal samples of symptomatic patients with suspected COVID-19 infection | Third week after inclusion
  Using IgG serological assay (EUROIMMUN Anti-SARS-Cov2 ELISA Ig) as gold/reference standard
To determine the ability of a clinical diagnosis based both on patients' symptoms and chest CT-scan to detect the SARS-CoV-2 in symptomatic patients with suspected COVID-19 infection | Third week after inclusion
  Using IgG serological assay (EUROIMMUN Anti-SARS-Cov2 ELISA Ig) as gold/reference standard
To determine the agreements between nasopharyngeal samples and oropharyngeal samples | At inclusion
  Using ddPCR and RT-qPCR assays
To determine the agreements between a clinical diagnosis and ddPCR and RT-qPCR assays | At inclusion
  Using ddPCR and RT-qPCR assays
To assess the 28-day mortality rate | Up to the follow-up end (28 days after inclusion)
  Rate calculated from the date of the first diagnostic procedure to the date of death of any cause
To determine potential predictive factors of death among patients' characteristics | Up to the follow-up end (28 days after inclusion)
  Demographics, type of tumor, type of anticancer, treatment, comorbidities, biological parameters
To evaluate the over risk of death of patients COVID+ versus COVID- | Up to the follow-up end (28 days after inclusion)
  After adjusting on main clinical characteristics and treatment type

OTHER OUTCOMES:
To evaluate the sensibility, specificity and diagnostic accuracy of "in-house" serologic test for the SARS-CoV-2 detection | At inclusion
  Comparison of our "in-house" test to the commercial serology test from EUROIMMUN used for the study

CONTACTS AND LOCATIONS:
Overall Officials: Bénédicte MASTROIANNI, MD, Principal Investigator — Centre Léon Berard
Locations (1):
- Centre Leon Berard, Lyon, France